CLINICAL TRIAL: NCT01566032
Title: Digital Versus Analog Pleural Drainage in Patients With Pulmonary Air Leak
Acronym: DiVA
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2011619-01H
Record Dates: First submitted 2012-03-26; First posted 2012-03-29 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Air Leak
Keywords: pulmonary air leak; Thopaz; analog; digital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The amount of air leaking from a chest tube can be measured in two main ways:

1. electronic monitor connected to the chest tube
2. numerical (non-electronic) monitor connected to the chest tube

For people who have had lung surgery, it is important to understand the impact of measuring air leaks accurately in both the short term and the long term. An electronic medical device called Thopaz measures air leak electronically. Another medical device called Pleur-evac measures air leak numerically. The purpose of this study is to understand the accuracy of the method used by doctors and nurses to determine if a chest tube has an air leak. It is also important to determine the size or severity of an air leak.

DETAILED DESCRIPTION:
Patients with air leaks following lung surgery will be assessed by a target number of 6 observers each (three nurses and three MDs) who will be randomly asked to participate. Patients will first be connected to the numerical air leak detector, followed by the electronic air leak detector. Observers will record their responses for each device. They will be blinded to responses from other observers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over
* Male and Female.
* Air leak occuring after any pulmonary resection
* Air leak persisting on or after the first post-op day of pleural drainage
* Air leak not entirely secondary to poor air seal at the pleural drainage incision site
* Pulmonary resection for benign or neoplastic diagnosis

Exclusion Criteria:

* Tension pneumothorax
* Traumatic or iatrogenic pneumothorax
* Primary or recurrent spontaneous pneumothorax awaiting surgery
* Pneumonectomy patient (history of or current)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A target of 30 patients at the Ottawa Hospital who experienced pulmonary air leak following pulmonary resection will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Inter-rater variability of air leak measurements. | Post-op
  Time frame will occur once patients have experienced an air leak. 70% of patients are expected to have a PAL on postoperative day 1. There will be a 4 hour window to complete observations from the numerical device. These observations will be followed by observations on digital device. Each observer should spend 5-10 min to complete both tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Gilbert, MD, Principal Investigator — Ottawa Hospital/Ottawa Hospital Research Institute
Locations (1):
- Ottawa General Hospital, Ottawa, Ontario, Canada